CLINICAL TRIAL: NCT03425279
Title: A Phase 1/2 Dose Escalation and Dose Expansion Study of Mecbotamab Vedotin (BA3011) Alone and in Combination With Nivolumab in Adult and Adolescent Patients 12 Years and Older With Advanced Solid Tumors
Brief Title: CAB-AXL-ADC Safety and Efficacy Study in Adult and Adolescent Patients With Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioAtla, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA3011-001
Record Dates: First submitted 2018-01-22; First posted 2018-02-07 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Undifferentiated Pleomorphic Sarcoma; Myxofibrosarcoma
Keywords: late stage; stage 3; stage 4; cancer; undifferentiated pleomorphic sarcoma; myxofibrosarcoma
MeSH Terms: conditions — Histiocytoma, Malignant Fibrous; Dermatofibrosarcoma; Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BA3011 (Experimental): Phase 1: All patients will receive BA3011, CAB-AXL-ADC.
  Phase 2: All patients will receive either BA3011 alone or in combination with PD-1 inhibitor.
  Interventions: Biological: CAB-AXL-ADC
- Combination Therapy (Experimental): Phase 2: BA3011 in combination with PD-1 inhibitor.
  Interventions: Biological: CAB-AXL-ADC; Biological: PD-1 inhibitor

INTERVENTIONS:
Biological: CAB-AXL-ADC — Conditionally active biologic anti-AXL antibody drug conjugate
Biological: PD-1 inhibitor — PD-1 inhibitor
  Arms: Combination Therapy

SUMMARY:
The objective of this study is to assess the safety and efficacy of mecbotamab vedotin (BA3011) in solid tumors.

DETAILED DESCRIPTION:
This is a multi-center, open-label, Phase 1/2 study designed to evaluate the safety, tolerability, PK, immunogenicity, and antitumor activity of mecbotamab vedotin (BA3011), a conditionally active biologic (CAB) AXL-targeted antibody drug conjugate (CAB-AXL-ADC) in patients with advanced solid tumors.

Phase 1 of this study will consist of a dose escalation phase (enrollment complete as of Oct 2019) and a dose expansion phase (enrollment complete as of Jan 2024).

Phase 2 will consist of two parts. Part 1 is designed to evaluate mecbotamab vedotin alone and with nivolumab in patients with various types of advanced sarcomas (enrollment complete as of Jan 2024). Part 2 will evaluate the safety and efficacy of mecbotamab vedotin in patients with undifferentiated pleomorphic sarcoma (UPS) and myxofibrosarcoma (MFS).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have measurable disease.
* Age ≥ 12 years (Phase 2)
* Adequate renal function
* Adequate liver function
* Adequate hematological function
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of at least three months.

Exclusion Criteria:

* Patients must not have clinically significant cardiac disease.
* Patients must not have known non-controlled CNS metastasis.
* Patients must not have a history of ≥ Grade 3 allergic reactions to mAb therapy as well as known or suspected allergy or intolerance to any agent given during this study.
* Patients must not have had major surgery within 4 weeks before first BA3011 administration.
* Patients must not have had prior therapy with a conjugated or unconjugated auristatin derivative/vinca-binding site targeting payload.
* Patients must not have known human immunodeficiency virus (HIV) infection, active hepatitis B and/or hepatitis C.
* Patients must not be women who are pregnant or breast feeding.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Phase 1: Safety Profile | Up to 24 months
  Assess dose limiting toxicity as defined in the protocol
Phase 1: Safety Profile | Up to 24 months
  Assess maximum tolerated dose as defined in the protocol
Phase 1 and 2: Safety Profile | Up to 24 months
  Frequency and severity of AEs and/or SAEs, and changes from baseline in laboratory parameters and vital signs
Phase 2: Confirmed overall response rate (ORR) per RECIST v1.1 | Up to 24 months
  Proportion of patients who achieve a confirmed CR or PR according to RECIST v1.1

SECONDARY OUTCOMES:
Phase 1: Pharmacokinetics | Up to 24 months
  Plasma concentrations of ADC, total antibody and MMAE
Phase 1: Pharmacokinetics | Up to 24 months
  Peak Plasma Concentration (Cmax)
Phase 1: Pharmacokinetics | Up to 24 months
  Area under the plasma concentration versus time curve (AUC)
Phase 1: Overall response rate (ORR) | Up to 24 months
  Proportion of patients who achieve a confirmed CR or PR
Phase 1: Immunogenicity | Up to 24 months
  The number and percentage of patients who develop detectable anti-drug antibodies (ADAs)
Phase 1 and 2: Duration of response (DOR) | Up to 24 months
  Time from the first documented OR until the first documented disease progression or death (due to any cause), whichever occurs first
Phase 1 and 2: Progression-free survival (PFS) | Up to 24 months
  Time from the first dose of IP until the first documentation of disease progression or death due to any cause, whichever occurs first
Phase 1 and 2: Best overall response (BOR) | Up to 24 months
  All post-baseline disease assessments that occur prior to the initiation of subsequent anticancer therapy
Phase 1 and 2: Disease control rate (DCR) | Up to 24 months
  Proportion of patients with a best overall response of confirmed CR, confirmed PR, or stable disease (SD) ≥ 12 weeks
Phase 1 and 2: Time to response (TTR) | Up to 24 months
  Time from the first dose of investigational product until the first documentation of OR
Phase 1 and 2: Overall survival (OS) | Up to 24 months
  Time from the first dose of BA3011 treatment until death due to any cause
Phase 1 and 2: Tumor size | Up to 24 months
  Percent change from baseline in tumor size

CONTACTS AND LOCATIONS:
Locations (40):
- United States (35):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Tower Hematology Oncology Medical Group, Los Angeles, California
  - Precision NextGen Oncology, Los Angeles, California
  - UCSF Medical Center - Cancer Immunotherapy Clinic (CIC), San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Sarah Cannon Research Institute at Health One, Denver, Colorado
  - Children's Research Institute, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Comprehensive Cancer Center of Nevada, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Abramson Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided